CLINICAL TRIAL: NCT06669494
Title: Analysis of Data and Development of Physical Function Assessment Indicators for Early Diagnosis and Monitoring Factors of Acquired Weakness in the Intensive Care Unit
Brief Title: Data Analysis and Physical Function Evaluation Index Development for Early Diagnosis and Monitoring of ICU-acquired Weakness
Acronym: Beyond ICU
Status: Enrolling by invitation | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health and Welfare (Ambiguous)
Responsible Party: Principal Investigator, Jong Geol Do, M.D, PhD, Assistant professor, Samsung Medical Center
Other Study IDs: 2024-06-107
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cohort Studies; ICU Acquired Weakness (ICUAW); Critical Illness
Keywords: Post Intensive Care Syndrome(PICS); Intensive Care Unit acquired weakness; Early mobilization; Digital Health Care Device
MeSH Terms: conditions — Critical Illness; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: This exploratory study aims to investigate the relationship between activity levels/muscle mass and clinical indicators. ., assuming an estimated Spearman's rank correlation of 0.7, a sample size of 43 participants would yield a two-sided 95% confidence interval with a margin of error of 0.17. Considering a dropout rate of 15%, a total of 51 participants is required.
  This study will begin enrolling ICU patients with weakness following approval from the Institutional Review Board (IRB). With an estimated enrollment rate of fewer than one participant per week, the enrollment period is expected to last approximately 12 months.
  -Lifelog via Wearable Device (Accelerometer::Fitbit) Participants will wear the Fitbit Charge 5 from the time of study registration after ICU admission until two weeks post-ICU discharge.
  If the participant meets the criteria for sarcopenia based on bioelectrical impedance analysis (BIA), a nerve conduction study will be conducted

SUMMARY:
Data Analysis and Physical Function Evaluation Index Development for Early Diagnosis and Monitoring of ICU-acquired weakness

DETAILED DESCRIPTION:
ICU-acquired weakness (ICU-AW) is a prevalent complication, occurring in more than 50% of ICU patients, and has severe long-term effects on patient outcomes. This condition not only prolongs the duration of hospital stay but also persists long after discharge, continuously impacting patients' health and quality of life. Therefore, monitoring, prevention, and rehabilitation of ICU-AW should not be limited to the ICU period but should continue after transfer to general wards and after discharge. This study aims to provide foundational data for developing a platform capable of continuously monitoring and delivering rehabilitation therapy for ICU-AW from ICU admission through the post-discharge period.

Recent meta-analyses have shown that providing rehabilitation for ICU patients improves physical function at discharge, reduces ICU stay by 0.8 days, and shortens total hospital stay by 1.75 days. Additionally, it increases the distance patients can walk unassisted at discharge, the number of patients capable of standing, the duration of ventilator-free days, and the percentage of patients discharged home. Understanding the recovery process of ICU-AW as a continuum from ICU to post-discharge is essential, and the necessity of continuous rehabilitation throughout this process is evident. However, the challenge lies in implementing this in real-world practice.

This study seeks to provide foundational data for developing personalized educational programs applicable to remote digital therapeutics in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU who are 19 years of age
* Patients who did consent of the study

Exclusion Criteria:

* Patients with a history of peripheral nerve injury
* Patients with a history of major surgery within the past 12 weeks or those expected to undergo major surgery during the trial period
* Patients with a history of central nervous system disorders (e.g., stroke, spinal cord injury)
* Patients with cognitive impairment that may interfere with the conduct of the study
* Patients with Do Not Resuscitate (DNR) orders, brain lesions, Clinical Frailty Score (CFS) exceeding 4, or those who have undergone cardiopulmonary resuscitation
* Patients confirmed to have metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the MICU who are 19 years of age, SamsungMC
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
MRC sum | Within 72 hours of ICU admission
  Total Score 60, 12-group muscles, each score 0-5. The Score below 48 is diagnosed a s ICU aquired weakness.
Grip strength | Within 72 hours of ICU admission
  To assess forearm strength, grip strength is measured using a dynamometer. Two measurements are taken on both the left and right sides, and the average value is recorded.
FSS-ICU | Within 72 hours of ICU admission
  Functional status Score for the4 Intensive Care Unit 5 Functional movement : Rolling / Supine to Sit / Sit to Stand / Sitting on the edge of the bed, Walking Each item is scored from 0 to 7 based on the level of assistance needed, with 0 indicating complete inability and 35 indicating independent function.
JH-highest mobility scale | Within 72 hours of ICU admission
  There are a total of 8 stages :
  lying in bed(1pt) Limited to activities in bed only(2 pt) Sitting up in bed (3 pt) Sitting on a chair beside the bed(4 pt) Standing(5 pt) Walking 10 steps beside the bed(6pt) Walking more than 7 meters (7pt) Walking more than 76 meters (8 pt)
Body composition | Within 72 hours of ICU admission
  Height, weight, BMI, body fat percentage, Muscle mass are measured using an InBody device
US ( muscle thickness) | Within 72 hours of ICU admission
  Muscle Thickness for a total of 6 tems in the upper and lower limbs, swallowing muscles , is measured using ultrasound examination
Fitbit charge 5 | During ICU status
  Activity amount assessment The Fitbit Charge 5 is a wristband device equipped with an accelerometer that detects movement across three axes. It tracks information such as step count, distance traveled, calories burned, and active minutes, recording data from the time of wear until the battery depletes. This wearable device enables lifelogging through accelerometry. The Fitbit Charge 5 will be worn continuously from ICU admission upon study enrollment through to two weeks post-ICU discharge.
Nerve conduction study | Within 72 hours of ICU admission
  IF Sarcopenia are met via Body Composition Assessment, nerve conduction study (NCS) is performed. NCS is conducted to evaluate peripheral nerve function and to determine the presence of peripheral neuropathy in this study. The nerve conduction study uses electrical stimulation to measure nerve conduction velocity, latency, and amplitude
Clinical Characteristics | Within 72 hours of ICU admission
  Age,Diagnosis,CCI,Medical History,Education Level,Marital status

SECONDARY OUTCOMES:
MRC sum | Within 24 hours of ICU discharge
  Total Score 60, 12-group muscles, each score 0-5. The Score below 48 is diagnosed a s ICU aquired weakness.
Grip strength | Within 24 hours of ICU admission
  To assess forearm strength, grip strength is measured using a dynamometer. Two measurements are taken on both the left and right sides, and the average value is recorded.
FSS-ICU | Within 24 hours of ICU discharge
  Functional status Score for the4 Intensive Care Unit 5 Functional movement : Rolling / Supine to Sit / Sit to Stand / Sitting on the edge of the bed, Walking Each item is scored from 0 to 7 based on the level of assistance needed, with 0 indicating complete inability and 35 indicating independent function.
JH-highest mobility scale | Within 24 hours of ICU discharge
  There are a total of 8 stages :
  lying in bed(1pt) Limited to activities in bed only(2 pt) Sitting up in bed (3 pt) Sitting on a chair beside the bed(4 pt) Standing(5 pt) Walking 10 steps beside the bed(6pt) Walking more than 7 meters (7pt) Walking more than 76 meters (8 pt)
Fitbit charge 5 | Within 24 hours of ICU discharge
  Activity amount assessment The Fitbit Charge 5 is a wristband device equipped with an accelerometer that detects movement across three axes. It tracks information such as step count, distance traveled, calories burned, and active minutes, recording data from the time of wear until the battery depletes. This wearable device enables lifelogging through accelerometry. The Fitbit Charge 5 will be worn continuously from ICU admission upon study enrollment through to two weeks post-ICU discharge.
US -muscle thickness (T2) | Within 24 hours of ICU discharge
  Muscle Thickness for a total of 6 tems in the upper and lower limbs, swallowing muscles , is measured using ultrasound examination
Body composition(T2) | Within 24 hours of ICU discharge
  Height, weight, BMI, body fat percentage, Muscle mass are measured using an InBody device

OTHER OUTCOMES:
JH-highest mobility scale(T3) | After 2 weeks of GW admission
  There are a total of 8 stages :
  lying in bed(1pt) Limited to activities in bed only(2 pt) Sitting up in bed (3 pt) Sitting on a chair beside the bed(4 pt) Standing(5 pt) Walking 10 steps beside the bed(6pt) Walking more than 7 meters (7pt) Walking more than 76 meters (8 pt)
MRC sum (T3) | After 2 weeks of GW admission
  Total Score 60, 12-group muscles, each score 0-5. The Score below 48 is diagnosed a s ICU aquired weakness.
Fitbit charge 5 (T3) | After 2 weeks of GW admission
  Activity amount assessment The Fitbit Charge 5 is a wristband device equipped with an accelerometer that detects movement across three axes. It tracks information such as step count, distance traveled, calories burned, and active minutes, recording data from the time of wear until the battery depletes. This wearable device enables lifelogging through accelerometry. The Fitbit Charge 5 will be worn continuously from ICU admission upon study enrollment through to two weeks post-ICU discharge.
FSS-ICU(T3) | After 2 weeks of GW admission
  Functional status Score for the4 Intensive Care Unit 5 Functional movement : Rolling / Supine to Sit / Sit to Stand / Sitting on the edge of the bed, Walking Each item is scored from 0 to 7 based on the level of assistance needed, with 0 indicating complete inability and 35 indicating independent function.
Grip strength(T3) | After 2 weeks of GW admission
  To assess forearm strength, grip strength is measured using a dynamometer. Two measurements are taken on both the left and right sides, and the average value is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Registration number, age, gender, study measurements.
Supporting Information: Study Protocol
Time Frame: From October 1, 2025, to October 1, 2028.